CLINICAL TRIAL: NCT04602949
Title: Detection of the 2019 Novel Coronavirus (SARS-CoV-2) Using Breath Analysis - Validation Study
Brief Title: Detection of COVID-19 Using Breath Analysis - Validation Study
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scentech Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Cov-2-SMC-2020
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2022-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 patients (Experimental): subjects who were found as COVID-19 positive patients by swab RT-PCR
  Interventions: Diagnostic Test: Breath Biopsy Analysis
- Healthy controls (Other): subjects who were found as COVID-19 Negative, by swab RT-PCR
  Interventions: Diagnostic Test: Breath Biopsy Analysis

INTERVENTIONS:
Diagnostic Test: Breath Biopsy Analysis — Analysis of a single breath Biopsy

SUMMARY:
DETECTION OF THE 2019 NOVEL CORONAVIRUS (SARS-CoV-2) USING BREATH ANALYSIS- VALIDATION STUDY

DETAILED DESCRIPTION:
A diagnostic prospective single-site study, with no anticipated risks or constraints.

Primary objective- To validate the value of a set of breath VOC biomarkers that enable us to distinguish between Coronavirus (SARS-CoV-2) carriers and SARS-CoV-2-negative in comparison to the gold-standard testing methodology.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 75 years at the time of consent
* Capable of understanding written and/or spoken language
* Able to provide informed consent
* Was not treated with Anti-viral drugs

Exclusion Criteria:

* Age under 6 years old
* Under guardianship or deprived of liberty
* Pregnant or lactating woman

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2558 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Presence of Volatile Organic Compounds indicating carriers of COVID-19. | Through the study completion, up to 3 months.
  Comparison of Volatile Organic Compounds found among COVID-19 carriers and Healthy controls.

SECONDARY OUTCOMES:
Association of exhaled biomarkers with participants' characteristics (age, gender, symptoms-severity, etc.). | Through the study completion, up to 3 months.
  Correlation level between exhaled biomarkers and participants' demographic characteristics.
sensitivity level of biomarkers' algorithm. | Through the study completion, up to 3 months.
  comparison of algorithm's sensitivity level to the sensitivity of COVID-19 swab TEST.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Dror, PhD, Study Director — Scentech Medical Technologies Ltd
Locations (1):
- Shamir Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No
No IPD is to be shared with other researchers.